CLINICAL TRIAL: NCT00482365
Title: A National Registry of Patients With Hepatocellular Carcinoma
Brief Title: National Registry and Blood Bank of Patients With Liver Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Sunil K. Geevarghese, Assistant Professor of Surgery; Director, Transplant Center Clinical Trials Office; Director, Living Donor Transplant Program; Liver and Hepatobiliary Surgeon, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC GI 0224; VU-VICC-GI-0224; VU-VICC-IRB-020116
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-05

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: biologic sample preservation procedure — biologic sample preservation procedure
  Other Names: blood draw and storage
Other: medical chart review — review of patients' medical records at study entry and every 6 months
Other: Patient interview — Elicit demographic data as well as information about personal habits such as drinking and smoking.

SUMMARY:
RATIONALE: Gathering health information about patients with liver cancer over time may help doctors learn more about the disease and may help the study of cancer in the future.

PURPOSE: This clinical trial is developing a national registry and blood bank of patients with liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate etiologic factors associated with hepatocellular carcinoma (HCC) in different ethnic groups and in different parts of the United States by developing a national registry of HCC patients.
* Survey stage and potential treatability of HCC patients referred to Vanderbilt University Hospital.
* Establish a serum repository for registry patients with samples to be used for future studies of the pathogenesis of chronic liver disease and HCC and for developing better diagnostic tests.

OUTLINE: This is a multicenter, cross-sectional database study.

Data are collected on patients diagnosed with hepatocellular carcinoma at Vanderbilt University Medical Center and at other participating hospitals or liver transplantation centers around the country for inclusion in a national registry of liver cancer patients. Registry data are collected at baseline and then every 6 months for up to 5 years. The data are derived from investigator interviews with patients and from medical chart review of routine medical care provided during the course of the study. Data are collected from all study sites and entered into a master database that includes information on patient demographics, diagnoses and staging details, treatment history, results of laboratory studies, and patient outcomes. Information derived from the registry is available to investigators at all study sites.

Patients in the registry also undergo blood collection at baseline. Blood samples are stored in a serum repository for evaluation in future studies related to liver disease, viral hepatitis, and liver cancer. A biological marker that may be analyzed is squamous cell carcinoma antigen immune complex (SCCA-IC).

PROJECTED ACCRUAL: A total of 1,500 patients will be accrued for the Vanderbilt University Medical Center study and up to 2,000 patients for the national study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatocellular carcinoma at a participating institution

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified as having Hepatocellular carcinoma (HCC).
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2002-04; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Etiologic factors associated with hepatocellular carcinoma in different ethnic groups across the US | every 6 months up to 5 years
  A descriptive analysis will be done to describe the number of patients with HCC, their underlying etiology, correlation between etiology and demographic features and the outcome of various forms of therapy. Survival analysis will be done, comparing various forms of therapy while adjusting for stage of disease.

SECONDARY OUTCOMES:
Serum repository for registry patients | At study entry
  blood samples will be drawn at the time of standard of care and stored.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Geevarghese, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee